CLINICAL TRIAL: NCT01845298
Title: Immune Activation and Drug Absorption in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TMC114HIV4076
Record Dates: First submitted 2013-04-29; First posted 2013-05-03 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Rifampin; rifamycin SV

ARMS (1):
- HIV-infected subjects (Experimental): HIV-infected subjects who have not yet initiated highly active antiretroviral therapy (HAART). All enrolled subjects will receive a single dose of rifampicin 600 mg.
  Interventions: Drug: Rifampicin 600 mg

INTERVENTIONS:
Drug: Rifampicin 600 mg — The investigators will administer a single dose of rifampicin 600 mg to study subjects in order to conduct a pharmacokinetic study of rifampicin absorption.
  Other Names: rifamycin

SUMMARY:
The investigators' objective is to describe the variability of rifampicin absorption, markers of inflammation and gut damage, intestinal absorptive capacity, and intestinal permeability among HIV-infected volunteers. Rifampicin is the least well absorbed of the first-line anti-tuberculosis drugs. Rifampicin malabsorption is frequently observed in HIV-infected patients with active tuberculosis, but cannot be predicted by patient factors such as CD4+ T cell count, viral load, or the presence of diarrhea. The mechanisms for rifampicin malabsorption in HIV-infected patients are unknown. An understanding of mechanisms for rifampicin malabsorption could eventually lead to new therapeutic targets, with the ultimate goal of improving HIV/tuberculosis treatment outcomes.

DETAILED DESCRIPTION:
The dosing scheme for rifampicin for the treatment of tuberculosis was developed in the pre-HIV era, and achieving target concentrations at the site of infection is important for a successful outcome. Rifampicin is the least well absorbed of the first-line anti-TB drugs and may depend on active transport across the intestinal barrier. Rifampicin malabsorption is frequently observed in HIV/tuberculosis patients, but cannot be predicted by patient factors such as CD4+ T cell count, viral load, or the presence of diarrhea. Most importantly, loss of rifampicin absorptive capacity in the setting of HIV infection would explain the inferior treatment outcomes that are characteristic of HIV-associated tuberculosis, including early mortality, relapse after the completion of therapy, and the development of rifampicin-resistant infection during anti-tuberculosis therapy.

The gut-associated lymphoid tissue is the site of early and dramatic lymphocyte depletion in HIV+ patients, with near complete loss of intestinal CCR5+ CD4+ T cells within the first few weeks of infection. Lymphocyte depletion is accompanied by the loss of intestinal epithelial barrier integrity, and recent attention has focused on potential role of bacterial translocation across the damaged ("leaky") intestinal barrier. In support of this model, systemic immune activation markers have been shown to predict HIV progression better than CD4+ T cell count or HIV viral load. Independent of the potential role of bacterial translocation, the damage to gut epithelium may have other profound consequences for the HIV-infected patient.

The impact of this disease progression on the enterocyte's capacity to absorb specific drugs and nutrients has not been adequately explored. Loss of rifampicin absorptive capacity in the setting of HIV infection would explain the inferior treatment outcomes that are characteristic of HIV-associated tuberculosis, including early mortality, relapse after the completion of therapy, and the development of rifampicin resistant infection during anti-tuberculosis therapy. Therefore, we propose a pilot study of the relationship between immune activation, rifampicin absorption, and intestinal capacity for carrier-mediated transport and permeability, which will lay the foundation for a K23 Career Development Award application to the Division of AIDS, NIAID.

Rifampicin is an-antibacterial compound from the rifamycin family that is used for the treatment of certain bacterial infections, and is the cornerstone of the first-line treatment regimen for tuberculosis. Polymorphisms in a specific drug uptake transporter gene, SLCO1B1, lead to significant variability in the pharmacokinetics of rifampicin. Other host factors that negatively influence rifampicin absorption are not well understood, particularly in the high-risk group of HIV-infected patients with active tuberculosis.

Long-term use of rifampicin is rarely associated with adverse effects that include a flu-like illness and anemia. Both of these effects cease after termination of the drug. Neither of these effects has been reported after a single dose administration. Hypersensitivity reactions presenting with rash have also been reported after prolonged use of rifampicin, but would be rare after a single-dose administration. The risks associated with rifampicin have been minimized by studying pharmacokinetics after administration of a single dose, rather than after prolonged use. Rifampicin is a potent inducer of the cytochrome p450 enzyme system that is involved in the metabolism of many commonly used therapeutic compounds. For this reason, we will exclude participants who are receiving any prescription medications with clinically significant drug-drug interactions with rifampicin.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected males and females, between the ages of 21 and 45 years.
* Naïve to antiretroviral therapy
* T cell count greater than 350 cells/mm3
* Body Mass Index (BMI) greater or equal to 19 and less than or equal to 33.
* Weight greater than 60 kilograms.
* Ability and willingness to provide informed consent.
* Ability to swallow oral medications

Exclusion Criteria:

* Breastfeeding.
* Allergy or sensitivity to rifampicin.
* Prior history of documented active tuberculosis infection.
* Receipt of any investigational therapy, chemotherapy, or immune modulatory agents within 42 days prior to study entry.
* The following laboratory values obtained within 42 days prior to study entry:

Hemoglobin < 12.0 g/dL; Females: Hemoglobin < 11.0 g/dL Platelet count < 100,000/mm3 AST, ALT, and bilirubin > 5x ULN An estimated creatinine clearance < 80 mL/min based on the Cockroft-Gault equation

* Positive blood test for latent tuberculosis infection (T-SPOT)
* Female participants of reproductive potential must have a negative serum or urine pregnancy test performed with 28 days prior to study entry.

"Female participants of reproductive potential" is defined as women who have reached menarche or who have not been post-menopausal for at least 24 consecutive months (i.e. who have had menses within the preceding 24 months) or who have not undergone surgical sterilization (e.g. hysterectomy, or bilateral oophorectomy or salpingectomy).

* Female participants of reproductive potential that are using oral contraceptive pills (OCPs) must be willing to use barrier precautions for contraception for at least 7 days following each study visit.
* Use of any of the following prescription medications within 30 days prior to study entry, which may have drug-drug interactions with rifampicin, including (but not limited to):

  * Anti-coagulants (warfarin)
  * Cardiac drugs (digoxin, quinidine, verapamil, nifedipine, metoprolol, atenolol, carvedilol)
  * Hypoglycemics (rosiglitazone, pioglitazone, glipizide, repaglinide)
  * Proton pump inhibitors (omeprazole, esomeprazole,
  * Immune modulators (tacrolimus, cyclosporine)
  * Corticosteroids (dexamethasone, prednisone, hydrocortisone)
  * H2 blockers (ranitidine, cimetidine)
  * HMG CoA reductase inhibitors (atorvastatin, pravastatin, simvastatin)
  * Benzodiazepines (alprazolam, diazepam, midazolam, triazolam)
  * CNS-acting drugs (amitriptyline, buproprion, clozapine, phenytoin)
* Evidence of current ongoing tobacco use, illicit drug use, or average alcohol use of greater than 2 drinks per day.
* Any illness that, in the opinion of the study investigator, might confound the results of the study, or pose an additional risk to the subject by his or her participation in the study.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2014-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03-14 (Actual)

PRIMARY OUTCOMES:
Rifampicin Absorption (Ka) | Baseline
  The investigators will perform a pharmacokinetic study to assess rifampicin absorption among study subjects. Pharmacokinetic modeling will be used to assess the absorption rate constant (Ka) for each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Vinnard, MD, Principal Investigator — Faculty
Locations (1):
- Drexel University College of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gurumurthy P, Ramachandran G, Hemanth Kumar AK, Rajasekaran S, Padmapriyadarsini C, Swaminathan S, Bhagavathy S, Venkatesan P, Sekar L, Mahilmaran A, Ravichandran N, Paramesh P. Decreased bioavailability of rifampin and other antituberculosis drugs in patients with advanced human immunodeficiency virus disease. Antimicrob Agents Chemother. 2004 Nov;48(11):4473-5. doi: 10.1128/AAC.48.11.4473-4475.2004. PMID 15504887
- [Background] Chigutsa E, Visser ME, Swart EC, Denti P, Pushpakom S, Egan D, Holford NH, Smith PJ, Maartens G, Owen A, McIlleron H. The SLCO1B1 rs4149032 polymorphism is highly prevalent in South Africans and is associated with reduced rifampin concentrations: dosing implications. Antimicrob Agents Chemother. 2011 Sep;55(9):4122-7. doi: 10.1128/AAC.01833-10. Epub 2011 Jun 27. PMID 21709081
- [Background] Sharpstone D, Neild P, Crane R, Taylor C, Hodgson C, Sherwood R, Gazzard B, Bjarnason I. Small intestinal transit, absorption, and permeability in patients with AIDS with and without diarrhoea. Gut. 1999 Jul;45(1):70-6. doi: 10.1136/gut.45.1.70. PMID 10369707
- [Derived] Vinnard C, Manley I, Scott B, Bernui M, Adams J, Varghese S, Zentner I, Kutzler MA. A Pilot Study of Immune Activation and Rifampin Absorption in HIV-Infected Patients without Tuberculosis Infection: A Short Report. Tuberc Res Treat. 2017;2017:2140974. doi: 10.1155/2017/2140974. Epub 2017 Dec 21. PMID 29430306